CLINICAL TRIAL: NCT01094964
Title: HYMN: A Randomized Controlled Phase III Trial Comparing Hyperthermia Plus Mitomycin to a Second Course of Bacillus Calmette-Guerin or Standard Therapy in Patients With Recurrence of Non-Muscle Invasive Bladder Cancer Following Induction or Maintenance Bacillus Calmette-Guerin Therapy
Brief Title: Hyperthermia and Mitomycin C, Bacillus Calmette-Guerin, or Standard Therapy as Second-Line Therapy in Treating Patients With Recurrent Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Research Campaign Clinical Trials Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CRC-TU-BL3010-HYMN; CDR0000668528 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN85785327; EUDRACT-2008-005428-99; EU-21015; UCL-08/0365; KYOWA-CRC-TU-BL3010-HYMN; MREC-09/H0717/56
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2010-03

CONDITIONS: Bladder Cancer
Keywords: recurrent bladder cancer; stage 0 bladder cancer; stage I bladder cancer; adenocarcinoma of the bladder; squamous cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Interferon-alpha; Epirubicin; Mitomycin; Diathermy

INTERVENTIONS:
Biological: BCG solution
Biological: recombinant interferon alfa
Drug: epirubicin hydrochloride
Drug: mitomycin C
Other: laboratory biomarker analysis
Procedure: hyperthermia treatment
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Hyperthermia therapy kills tumor cells by heating them to several degrees above normal body temperature. Drugs used in chemotherapy, such as mitomycin C and epirubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as bacillus calmette-guerin (BCG) and interferon alfa, may stimulate the immune system in different ways and stop tumor cells from growing. It is not yet known whether giving hyperthermia together with mitomycin C is more effective than giving BCG or standard therapy as second-line therapy in treating patients with recurrent bladder cancer.

PURPOSE: This randomized phase III trial is studying how well hyperthermia given together with mitomycin C works compared with BCG or standard therapy as second-line therapy in treating patients with recurrent bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether hyperthermia in combination with mitomycin C versus bacillus Calmette-Guerin (BCG) or standard therapy as second-line therapy is effective in patients with recurrent non-muscle invasive bladder cancer following induction or maintenance therapy with BCG.
* To compare disease-free survival time in all patients.
* To compare complete response rate at 3 months in patients with carcinoma in situ.

Secondary

* To compare progression-free survival, overall survival, safety and tolerability of treatments, quality of life, cost, and cost-effectiveness in these patients.
* To assess biomarkers of response to standard and investigational treatment.

OUTLINE: This is a multicenter study. Patients are stratified according to presence of carcinoma in situ (yes vs no), prior bacillus Calmette-Guérin (BCG) therapy (induction vs maintenance), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I (experimental): Patients receive intravesical mitomycin C over two 30-minute instillations per session, and bladder hyperthermia (42 +/-2°C) is delivered in combination with each instillation. The suspension is maintained in the bladder for up to 2 hours. Treatment repeats once a week for 6 weeks followed by a 6-week rest period. Patients who are disease-free proceed to maintenance therapy consisting of one instillation of mitomycin C with bladder hyperthermia every 6 weeks for 1 year and then once every 8 weeks for 1 year. Patients who are disease-free at 24 months may continue treatment at the discretion of the clinician.
* Arm II (control): Patients receive 1 of the following treatment regimens depending on prior BCG treatment.

  * Second course of BCG therapy (patients who failed previous induction BCG): Patients receive intravesical BCG (1 instillation) once a week for 6 weeks. The suspension is maintained in the bladder for up to 2 hours. Patients then receive maintenance therapy consisting of BCG once a week for 3 weeks in months 3, 6, 12, 18, and 24. Patients who are disease-free at 24 months may continue treatment at the discretion of the clinician.
  * Standard therapy (patients who failed previous maintenance BCG): Patients receive standard therapy for BCG failure as defined by their treating centers. Standard therapy may include intravesical BCG alone, intravesical mitomycin C alone, intravesical epirubicin hydrochloride alone, or intravesical BCG in combination with interferon alpha.

All patients undergo cystoscopic surveillance with or without a biopsy every 3 months for 2 years. Urine, blood, and tissue samples are collected periodically for biomarker laboratory studies. Patients complete quality of life questionnaires (EORTC QLQ-BLS24, QLQ-C30, and EQ5D) at baseline, at 12 weeks, and at 6, 9, and 12 months.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-muscle invasive bladder cancer
* Recurrent disease after undergoing induction or maintenance therapy with bacillus Calmette-Guérin (BCG), meeting any 1 of the following criteria:

  * Stage Ta or T1 disease (grade 2 or 3)
  * Carcinoma in situ with stage Ta or T1 disease (grade 1, 2, or 3)
  * Carcinoma in situ alone
* Has undergone a second resection of all T1 disease to exclude muscle invasive disease
* No urothelial cell carcinoma (UCC) ≥ T2
* No recurrence of grade 1 UCC following BCG induction therapy
* No UCC involving the prostatic urethra or upper urinary tract

PATIENT CHARACTERISTICS:

* WHO performance status 0-4
* WBC ≥ 3.0 x 10^9/L
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100 x 10^9/L
* Serum creatinine < 1.5 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Normal kidneys and ureters on imaging CT scan within the past 12 months
* Available for long-term follow-up with a life expectancy of the duration of the trial
* Must be fit and willing to undergo a full or partial cystectomy
* No known or suspected reduced bladder capacity (< 250 mL)
* No significant bleeding disorder
* No other malignancy within the past 5 years except nonmelanomatous skin cancer cured by excision, adequately treated carcinoma in situ of the cervix, or DCIS/LCIS of the breast
* No known allergy to mitomycin or bacillus Calmette-Guérin (BCG), or previously withdrawn from BCG treatment due to a related adverse event (e.g., systemic infection)
* No active or intractable urinary tract infection
* No urethral stricture or any situation impeding the insertion of a 20F catheter
* No bladder diverticula > 1 cm
* No significant urinary incontinence
* No concurrent implanted electronic devices (e.g., cardiac pacemakers) or metallic implants within the pelvis, lower torso, spine, hip, or upper femur
* No immunocompromised state for any reason

PRIOR CONCURRENT THERAPY:

* At least 6 months since prior intravesical chemotherapy, except for single instillation post-transurethral resection
* No prior pelvic irradiation
* No prior hyperthermia in combination with intravesical mitomycin
* Concurrent participation in other studies allowed
* No current or long-term use of corticosteroids
* No concurrent chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time
Complete response rate at 3 months in patients with carcinoma in situ

SECONDARY OUTCOMES:
Recurrence-free survival time
Progression-free survival time
Overall survival time
Disease-specific survival time
Safety and tolerability
Quality of Life
Cost effectiveness
Biomarkers of response to standard and investigational treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Kelly, MD, Principal Investigator — University College London Hospitals
Locations (9):
- United Kingdom (9):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - University Hospitals of Leicester NHS Trust, Leicester, England
  - St. George's Hospital, London, England
  - University College of London Hospitals, London, England
  - South Manchester University Hospital, Manchester, England
  - James Cook University Hospital, Middlesbrough, England
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Derived] Tan WS, Panchal A, Buckley L, Devall AJ, Loubiere LS, Pope AM, Feneley MR, Cresswell J, Issa R, Mostafid H, Madaan S, Bhatt R, McGrath J, Sangar V, Griffiths TRL, Page T, Hodgson D, Datta SN, Billingham LJ, Kelly JD. Radiofrequency-induced Thermo-chemotherapy Effect Versus a Second Course of Bacillus Calmette-Guerin or Institutional Standard in Patients with Recurrence of Non-muscle-invasive Bladder Cancer Following Induction or Maintenance Bacillus Calmette-Guerin Therapy (HYMN): A Phase III, Open-label, Randomised Controlled Trial. Eur Urol. 2019 Jan;75(1):63-71. doi: 10.1016/j.eururo.2018.09.005. Epub 2018 Sep 28. PMID 30274699